CLINICAL TRIAL: NCT04505332
Title: Investigation of the Relationship Between Back Pain and Arthroplasty in Orthopedists
Brief Title: Back Pain and Arthroplasty in Orthopedists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ali Erkan YENİGUL, Principal Investigator, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.12.07
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Pain, Chronic; Back Pain
MeSH Terms: conditions — Chronic Pain; Back Pain | interventions — Arthroplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orthopedists (Other): orthopedists working actively and performing arthroplasty every day
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — back pain in orthopedists due to working actively and performing arthroplasty every day
  Other Names: back pain

SUMMARY:
The relationship between arthroplasty and low back pain in orthopedists will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Those who have received specialization of orthopaedics and work as a orthopaedics surgery.
* Those who want to participate in the study

Exclusion Criteria:

* Patients with discomfort and operation due to the low back pain
* Physicians in other branches

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
back pain in orthopedists | 2 month
  The relationship between arthroplasty performing and back pain in orthopaedics. Some orthopaedics perform arthroplasty every day, some perform 2 or 3 times a day. This can cause some pain in the low back due to the position during the operation. In our study, the investigators will have a survey of orthopaedics and answer some questions: How long have they been doing this job, how many arthroplasty operation they made during a day, do they have any complaints of low back pain. The investigators will try to relate back pain with their answers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Erkan YENIGUL, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No